CLINICAL TRIAL: NCT00385853
Title: A Phase I Study of PRK787/ZK 222584 in Combination With Daily Temozolomide and Radiation in Patients With Newly Diagnosed Glioblastoma
Brief Title: PTK787/ZK 222584 in Combination With Temozolomide and Radiation in Patients With Glioblastoma Taking Enzyme-Inducing Anti-Epileptic Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Tracy T. Batchelor, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-013
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Glioblastoma
Keywords: PTK; temozolomide; glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — vatalanib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTK787 (Experimental): Single arm study of PTK787
  Interventions: Drug: PTK787/ZK 222584; Drug: Temozolomide; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: PTK787/ZK 222584 — Twice daily for each 28-day cycle
Drug: Temozolomide — Daily for each 28-day cycle
Procedure: Radiation Therapy — For 7 weeks beginning on day 5 of the first treatment cycle

SUMMARY:
PTK is an investigational new drug that has been shown in early laboratory studies to prevent the formation of new blood vessels that allow the tumor to grow. These studies have shown that the study drug can potentially improve the effectiveness of additional radiation and chemotherapy. With this study, we would like to examine the effects of PTK when used in combination with radiation therapy and the anti-cancer drug temozolomide, the standard treatment for patients with newly diagnosed glioblastoma. We would also like to learn how the study drug is absorbed, distributed, and cleared from the body.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of PTK that can be administered safely without severe or unmanageable side effects, not everyone who participates will get the same dose of PTK. A small group will be enrolled onto the study and given a certain dose. If they tolerate it well, the next small group enrolled will receive a higher dose. This will continue until the highest dose that can be given without severe or unmanageable side effects is found.
* Participants will receive PTK twice daily along with temozolomide daily during each treatment cycle. Each treatment cycle lasts 28 days.
* PTK will start on Day 0 of the first cycle and will be given twice daily for the 7 weeks the participant receives radiation therapy.
* Daily doses of temozolomide will begin on Day of the first cycle and continue until the last dose of radiation therapy in cycle 1.
* Each participant will receive 7 weeks of radiation therapy. Radiation therapy will start on Day 5 of the first cycle and will be administered monday through friday, except on holidays.
* When radiation stops, temozolomide and PTK will be given for a maximum of 6 post-radiation cycles of study treatment. During these cycles, PTK and temozolomide will be given for 5 consecutive days followed by 23 days of no drugs.
* Tests will be performed routinely throughout the study treatment and include; chest x-rays, blood tests, physical exams, urine tests and ECG.
* The following procedures will be performed at the end of the study or after the participants last dose of study medication; tumor assessment by MRI, routine blood draws, neurological/physical exam and, medical history review.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically verified glioblastoma. Patients mus have paraffin blocks of tumor that must be sent for analysis.
* 18 years of age or older
* Karnofsky Performance Status greater than or equal to 60
* Adequate laboratory values as described by the protocol
* Life expectancy of greater than 12 weeks
* Patient must be able to undergo serial MR imaging
* Patients must be on an enzyme-inducing anti-epileptic drug(s) as listed in the protocol
* No steroids or a stable dose of steroids for at least 5 days or a decreasing dose
* Mini-mental status examination of 15 or greater

Exclusion Criteria:

* Pregnant or breast-feeding women
* Concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* Prior chemotherapy or cranial radiation therapy for glioblastoma
* Prior biologic or immunotherapy less than 2 weeks prior to registration
* If the patient surgery is more than 16 days or less than 13 days from the start of PTK787/ZK 222854
* Prior therapy with anti-VEGF agents
* Pleural effusion or ascites that causes respiratory compromise
* Concurrent severe and/or uncontrolled medical conditions which could compromise participation is the study
* Impairment of gastrointestinal function or GI disease that may significantly alter the absorption of PTK787/ZK 222584
* Confirmed diagnosis of human immunodeficiency virus (IV)
* Patients who are taking therapeutic warfarin sodium or other anticoagulants or anti-platelet agents
* Patients requiring aprepitant, dolasetron, and tropisetron as antiemetics are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose, safety and feasibility of PTK787/ZK 222584 in combination with temozolomide and radiation in patients with newly diagnosed glioblastoma. | 2 years

SECONDARY OUTCOMES:
Determine the pharmacologic profile of PTK787/ZK 222584 in this patient population | 2 years
determine the overall survival of patients with recurrent GM treated with PTK787/ZK 222584, when combined with temozolomide and radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Gerstner ER, Eichler AF, Plotkin SR, Drappatz J, Doyle CL, Xu L, Duda DG, Wen PY, Jain RK, Batchelor TT. Phase I trial with biomarker studies of vatalanib (PTK787) in patients with newly diagnosed glioblastoma treated with enzyme inducing anti-epileptic drugs and standard radiation and temozolomide. J Neurooncol. 2011 Jun;103(2):325-32. doi: 10.1007/s11060-010-0390-7. Epub 2010 Sep 7. PMID 20821342